CLINICAL TRIAL: NCT00562926
Title: Single Nucleotide Polymorphism (SNP) in Schizophrenia and Schizophrenia Spectrum Disorders: a Population Association Analysis With Hong Kong Chinese
Status: Completed | Type: Observational
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Chinese University of Hong Kong (Other)
Other Study IDs: CREC-2004, 247; HARECCTR0500025
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizophrenia spectrum disorder
MeSH Terms: conditions — Schizophrenia | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Extraction of 10ml blood sample for extraction of genomic DNA using DNA purification kits

SUMMARY:
Gamma-aminobutyric acid (GABA) is the principal inhibitory neurotransmitter in the mammalian central nervous system. It is involved in a wide spectrum of physiological functions, from sleep and sedation to convulsions. A defect in neurotransmission involving GABA in schizophrenia was first propsed in early 1970s, based on neuropathologcial evidence, yet there is a lack of molecular genetic evidence.

Recently, we carried out a pilot study on a region of the GABA-A receptor β2 subunit gene on chromosome 5 and found significant association for single nucleotide polymorphisms (SNPs) in the gene sequence with occurrence of schizophrenia. The current proposal aims to validate this important finding and to conduct a thorough scanning of the complete gene sequences of the GABA-A receptor subunit genes in this chromosomal region, including the three major subunits α1, β2 and γ2. We shall collect samples from Hong Kong Chinese subjects for a case-control study using haplotype maps and comparing the SNP haplotype frequencies in the receptor genes, and hence examine whether these genes are in association with schizophrenia, or other schizophrenia-spectrum disorders, including Alzheimer's disease presenting with psychotic symptoms.

Based on the observation that patients suffering from the catatonic subtype of schizophrenia respond particularly well to benzodiazepines, which bind specifically to GABA-A receptors, we shall also perform data analysis in terms of correlating SNP association with schizophrenia subtypes. Association of GABA-A receptor genes with schizophrenia would be a major step forward to determining whether these genes are susceptibility genes for schizophrenia, thereby paving the way to more effective diagnosis and treatment for this debilitating disease.

ELIGIBILITY:
Inclusion Criteria:

(For patients:)

* Diagnosis of schizophrenia under DSM-IV guidelines.

Exclusion Criteria:

(For controls:)

* Subjects who are known to have blood transmitted disease.
* Past or current alcohol and /or substance abuse.
* Past or current major medical and neurological conditions.

(For patients:)

* As for controls, excepr 3. "neurological conditions" does not include schizophrenia.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2004-07; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dicky WS Chung, Dr, Principal Investigator — Department of Psychiatry, Tai Po Hospital
Locations (4):
- China (4):
  - NTE Cluster under HA, Hong Kong
  - Shatin Hospital, Hong Kong
  - Tai Po Hospital, Hong Kong
  - The Hong Kong University of Science and Technology, Hong Kong